CLINICAL TRIAL: NCT03977207
Title: A Randomized Controlled Trial of Thyroid Hormone Supplementation in Hemodialysis Patients
Acronym: THYROID-HD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Irvine (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Principal Investigator, Connie Rhee, Assistant Professor of Medicine and Public Health; Division of Nephrology and Hypertension, Department of Medicine, University of California, Irvine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 20195142
Record Dates: First submitted 2019-05-28; First posted 2019-06-06 (Actual); Last update posted 2025-09-08 (Actual); Status verified 2025-08

CONDITIONS: Thyroid; Functional Disturbance; Hypothyroidism; Hemodialysis
MeSH Terms: conditions — Thyroid Diseases; Hypothyroidism | interventions — Thyroxine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Levothyroxine (Experimental): Patients will be randomized to levothyroxine or placebo (similar in size, shape, and color to levothyroxine) via permuted blocks stratified by two TSH levels (>3.0-5.0 and 5.0-10.0mIU/L) to ensure treatment balance across TSH levels. The study medications will be prepared in pill form. In the treatment arm, initial L-T4 doses will be 25mcg vs. 50mcg among patients whose TSH is >3.0-5.0mIU/L vs. 5.0-10.0mIU/L, respectively. Patients in the placebo arm will receive an equivalent number of placebo pills daily depending upon TSH level.
  The intervention period is 24 weeks. Patients will undergo up to two subsequent dose titrations after 8- and 16-weeks of treatment, based on interim TSH measurements at these time points. Patients whose TSH levels are higher or lower than the therapeutic TSH target of 0.5-3.0mIU/L will undergo a dose adjustment (+/- 25mcg), while those whose TSH levels are in target range will continue the prior dose.
  Interventions: Drug: Levothyroxine Sodium
- Placebo (Placebo Comparator): Patients will be randomized to levothyroxine or placebo (similar in size, shape, and color to levothyroxine) via permuted blocks stratified by two TSH levels (>3.0-5.0 and 5.0-10.0mIU/L) to ensure treatment balance across TSH levels. The study medications will be prepared in pill form. In the treatment arm, initial L-T4 doses will be 25mcg vs. 50mcg among patients whose TSH is >3.0-5.0mIU/L vs. 5.0-10.0mIU/L, respectively. Patients in the placebo arm will receive an equivalent number of placebo pills daily depending upon TSH level.
  The intervention period is 24 weeks. Patients in the placebo arm will undergo an equivalent titration in placebo pills (as that of the experimental arm) after 8- and 16-weeks of treatment, based on interim TSH measurements at these time points.
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Levothyroxine Sodium — Thyroid hormone supplement
  Arms: Levothyroxine
Drug: Placebos — Placebo oral capsule
  Arms: Placebo

SUMMARY:
Hypothyroidism, defined by elevated thyrotropin (TSH) levels, is a common endocrine complication in chronic kidney disease patients, and prior evidence shows that higher TSH levels, even within the normal laboratory range, are strongly associated with impaired quality of life and cardiovascular disease in this population. Levothyroxine is one of the most frequently prescribed medications in chronic kidney disease, yet its efficacy and safety in these patients have not been well-studied. Hence, this study will investigate 1) whether levothyroxine improves patient-centered (e.g., health-related quality of life, physical performance, strength) and 2) cardiovascular (e.g., coronary artery calcification, endothelial function, systolic function) outcomes in dialysis patients, and 3) if thyroid hormone replacement exerts classic metabolic effects (i.e., changes in body fat and resting energy expenditure) in this population.

DETAILED DESCRIPTION:
Data spanning over three decades show that hypothyroidism is highly prevalent in the chronic kidney disease (CKD) population, affecting 25% of those receiving dialysis therapy. In the general population hypothyroidism, defined by elevated thyrotropin (TSH) levels, has been associated with impaired health-related quality of life (HRQOL) and cardiovascular (CV) morbidity and mortality, but until recently there was a paucity of data regarding its prognostic implications in CKD. Our research has been the first to show a link between high-normal TSH levels and worse HRQOL Short Form 36 scores in dialysis patients, particularly among subscales centered on physical health (e.g., physical function, energy/fatigue). Our studies have also advanced the field by showing that elevated TSH levels even within the "normal" range (>3.0mIU/L) are associated with heightened risk of CV disease and death across multiple dialysis cohorts. However, there remains considerable controversy as to 1) whether thyroid dysfunction is causally associated with adverse patient-centered and CV outcomes, and 2) if elevated TSH levels represent thyroid functional disease vs. non-thyroidal illness in CKD. While levothyroxine is one of the most commonly prescribed medications in CKD, little is known about its efficacy in this population.

To address these knowledge gaps, we propose to conduct a randomized double-blind placebo-controlled trial among 336 hemodialysis patients with high-normal or subclinical hypothyroid range serum TSH levels to determine the effects of 24 weeks (i.e., 6 months) of levothyroxine vs. placebo on 1) HRQOL Short Form 36 (SF36) Physical Component Score and 2) coronary artery calcifcation (CAC) progression (co-primary endpoints).

As secondary endpoints, we will also examine 1) HRQOL measured by the ThyPRO survey, 2) physical performance, 3) endothelial function, 4) vascular calcification inhibitor levels, and 5) total body fat percentage. In a sub-study of 108 hemodialysis patients, we will also examine exploratory secondary endpoints of 1) muscle strength, 2) systolic function, and 3) resting energy expenditure.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-75 years old
* Received hemodialysis at least four weeks
* Have two consecutive thyrotropin (TSH) levels >3.0-10.0mIU/L during the screening period
* Have normal free thyroxine (FT4) levels
* Have ability to provide written informed consent

Exclusion Criteria:

* Active treatment with thyroid hormone supplementation or anti-thyroid medications
* Active receipt of dialysis
* Prior kidney transplantation
* Life expectancy less than six months
* Active malignancy or prior thyroid malignancy
* Active pregnancy or planning a pregnancy
* Active coronary ischemia or atrial fibrillation (evaluated by EKG)
* Active congestive heart failure exacerbation
* Osteoporosis
* Weight in excess of 450 lbs.
* Hyperthyroidism as determined by TSH <0.5mIU/L during the screening period, anti-thyroid medication use, or hyperthyroidism diagnosis

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 336 (Estimated)
Dates: Start 2020-07-20 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Health-Related Quality of Life (HRQOL) - Short Form 36 Physical Component Score | Week 0 (pre-trial/baseline)
  We will assess HRQOL using the Short Form 36, which consists of 36 questions grouped into eight subscales (score 0-100 for each subscale; higher scores indicate better states of health) that will be used to derive a summary Physical Component Score.
Health-Related Quality of Life (HRQOL) - Short Form 36 Physical Component Score | Week 12
  We will assess HRQOL using the Short Form 36, which consists of 36 questions grouped into eight subscales (score 0-100 for each subscale; higher scores indicate better states of health) that will be used to derive a summary Physical Component Score.
Health-Related Quality of Life (HRQOL) - Short Form 36 Physical Component Score | Week 24
  We will assess HRQOL using the Short Form 36, which consists of 36 questions grouped into eight subscales (score 0-100 for each subscale; higher scores indicate better states of health) that will be used to derive a summary Physical Component Score.
Coronary Artery Calcification (CAC) - Volume Score | Week 0 (pre-trial/baseline)
  We will assess CAC Volume Score using a 256-multidetector CT test. Volume score will be calculated by multiplying the number of voxels with calcification by the volume of each voxel for each calcified lesion, and summing individual lesion scores from the four main coronary arteries (left main, left anterior descending, circumflex, and right coronary artery).
Coronary Artery Calcification (CAC) - Volume Score | Week 24
  We will assess CAC Volume Score using a 256-multidetector CT test. Volume score will be calculated by multiplying the number of voxels with calcification by the volume of each voxel for each calcified lesion, and summing individual lesion scores from the four main coronary arteries (left main, left anterior descending, circumflex, and right coronary artery).

SECONDARY OUTCOMES:
Thyroid-Specific HRQOL - ThyPRO Hypothyroid Symptoms and Tiredness Domain Scores | Weeks 0 (pre-trial/baseline) and 24 (post-randomization)
  We will administer the thyroid-specific quality of life patient-reported outcome (ThyPRO) measure, which is comprised of 84 items categorized into 13 domains, plus a general quality of life question (this is a composite measure).
Physical Performance - Short Physical Performance Battery (SPPB) | Weeks 0 (pre-trial/baseline) and 24 (post-randomization)
  We will measure physical performance using the Short Physical Performance Battery (SPPB), which tests 1) gait speed (faster of two timed, usual pace 15-foot walks), 2) balance (balance test measuring ability to stand with feet in side-by-side, semi-tandem, and tandem positions for 10 seconds), and 3) chair raises (timed series of five attempts to arise from a chair unassisted without use of arms), with each component ranging from 0 to 4 (score 0-12; higher score indicates better performance).
Endothelial Function - Digital Thermal Monitor | Weeks 0 (pre-trial/baseline) and 24 (post-randomization)
  We will measure endothelial function using digital thermal monitor (DTM) testing, which is based on the principle that changes in fingertip temperature during and after an ischemic stimulus (blood pressure [BP] cuff occlusion) reflect changes in blood flow. In normal endothelial function, cuff inflation results in a 1-3 degree Celsius temperature decline, followed by rapid temperature rise to above baseline during cuff deflation due to compensatory vasodilation. Temperature (temp) will be measured before, during, and after a 2-minute BP cuff inflation in the non-vascular access arm in order to measure Area Under the Temp Curve (TMP-AUC), defined as area under the curve between the maximum and minimum temp.
Vascular Calcification Inhibitor - Matrix Gla Protein Levels | Weeks 0 (pre-trial/baseline) and 24 (post-randomization)
  We will use plasma collected during hemodialysis treatments to measure total uncarboxylated matrix Gla protein levels. Assays will be conducted in the University of California Irvine Institute of Clinical Translational Science Bioassay Core.
Total Body Fat Percentage | Weeks 0 (pre-trial/baseline) and 24 (post-randomization)
  We will assess total body fat percentage using Dual Energy X-Ray absorptiometry.
Muscle Strength - Isometric Dynamometry | Weeks 0 (pre-trial/baseline) and 24 (post-randomization)
  We will assess muscle strength using BioDex dynamometry, which will be used to measure Isometric Quadriceps Maximal Strength (Peak Torque, Newton-meters), in which patients will perform three maximal knee-extension efforts at a knee angle of 60 degrees using the dominant leg; each trial consists of a repetition of five seconds of concentric quadriceps contraction, followed by at least 90-seconds of resting recovery.
Systolic Function - Global Longitudinal Strain | Weeks 0 (pre-trial/baseline) and 24 (post-randomization)
  We will measure systolic function using Global Longitudinal Strain (GLS) using speckle-tracking 2D-echocardiography, which measures the contraction/deformation of myocardium during systole and is represented by a negative value (i.e., more negative GLS indicates better function).
Resting Energy Expenditure (REE) - Indirect Calorimetry | Weeks 0 (pre-trial/baseline) and 24 (post-randomization)
  We will measure REE using indirect calorimetry, in which following an overnight fast, patients will undergo a 20-minute resting period, after which oxygen consumption and carbon dioxide expiration will be recorded for 20-minutes while remaining under resting conditions, which will be used to calculate REE using the Weir formula.

CONTACTS AND LOCATIONS:
Locations (1):
- University of California Irvine, Orange, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rhee CM, Chen Y, You AS, Brunelli SM, Kovesdy CP, Budoff MJ, Brent GA, Kalantar-Zadeh K, Nguyen DV. Thyroid Status, Quality of Life, and Mental Health in Patients on Hemodialysis. Clin J Am Soc Nephrol. 2017 Aug 7;12(8):1274-1283. doi: 10.2215/CJN.13211216. Epub 2017 Jul 13. PMID 28705886
- [Background] Rhee CM, You AS, Nguyen DV, Brunelli SM, Budoff MJ, Streja E, Nakata T, Kovesdy CP, Brent GA, Kalantar-Zadeh K. Thyroid Status and Mortality in a Prospective Hemodialysis Cohort. J Clin Endocrinol Metab. 2017 May 1;102(5):1568-1577. doi: 10.1210/jc.2016-3616. PMID 28324018
- [Background] Rhee CM, Kim S, Gillen DL, Oztan T, Wang J, Mehrotra R, Kuttykrishnan S, Nguyen DV, Brunelli SM, Kovesdy CP, Brent GA, Kalantar-Zadeh K. Association of thyroid functional disease with mortality in a national cohort of incident hemodialysis patients. J Clin Endocrinol Metab. 2015 Apr;100(4):1386-95. doi: 10.1210/jc.2014-4311. Epub 2015 Jan 29. PMID 25632971
- [Background] Rhee CM, Alexander EK, Bhan I, Brunelli SM. Hypothyroidism and mortality among dialysis patients. Clin J Am Soc Nephrol. 2013 Apr;8(4):593-601. doi: 10.2215/CJN.06920712. Epub 2012 Dec 20. PMID 23258793
- [Background] Rhee CM, Ravel VA, Streja E, Mehrotra R, Kim S, Wang J, Nguyen DV, Kovesdy CP, Brent GA, Kalantar-Zadeh K. Thyroid Functional Disease and Mortality in a National Peritoneal Dialysis Cohort. J Clin Endocrinol Metab. 2016 Nov;101(11):4054-4061. doi: 10.1210/jc.2016-1691. Epub 2016 Aug 15. PMID 27525529
- [Background] Rhee CM, Kalantar-Zadeh K, Ravel V, Streja E, You AS, Brunelli SM, Nguyen DV, Brent GA, Kovesdy CP. Thyroid Status and Death Risk in US Veterans With Chronic Kidney Disease. Mayo Clin Proc. 2018 May;93(5):573-585. doi: 10.1016/j.mayocp.2018.01.024. PMID 29728200